CLINICAL TRIAL: NCT01167582
Title: Myocardial Ischemia and Transfusion Pilot
Acronym: MINT Pilot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Pittsburgh (Other); Albert Einstein College of Medicine (Other); Brigham and Women's Hospital (Other); Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey L Carson, MD, Jeffrey L Carson, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0220090205; 1RC2HL101458-01 (NIH)
Record Dates: First submitted 2010-03-17; First posted 2010-07-22 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Myocardial Infarction; Unstable Angina; Coronary Artery Disease
Keywords: blood transfusion; red blood cell transfusion; myocardial infarction; acute coronary syndrome; anemia
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable; Coronary Artery Disease; Acute Coronary Syndrome; Anemia | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal Transfusion Strategy (Experimental): Patients randomly allocated to the liberal transfusion strategy receive one unit of packed red cells following randomization and receive enough blood to raise the hemoglobin concentration above 10 g/dL any time the hemoglobin concentration is detected to be below 10g/dL during the hospitalization for up to 30 days. Any transfusion following the initial unit of packed red cells must be preceded by blood test documenting a hemoglobin concentration below 10 g/dL.
  Interventions: Biological: Red blood cell transfusion
- Restrictive transfusion strategy (Experimental): Receive a transfusion if they develop symptoms related to anemia. Transfusion is also permitted, but not required, in the absence of symptoms only if the hemoglobin concentration falls below 8 g/dL. Blood is administered one unit at a time and the presence of symptoms is reassessed. Only enough blood is given to relieve symptoms. If the transfusion is given because the hemoglobin concentration falls below 8 g/dL, then only enough blood is given to increase the hemoglobin concentration above 8 g/dL.
  Symptoms of anemia that will be indications for transfusion are: 1) Definite angina requiring treatment with sublingual nitroglycerin or equivalent therapy. 2) Unexplained tachycardia or hypotension.
  Interventions: Biological: Red blood cell transfusion

INTERVENTIONS:
Biological: Red blood cell transfusion — Liberal versus restrictive transfusion

SUMMARY:
The purpose of this study is to evaluate two approaches to red blood cell transfusion in anemic patients with acute coronary syndrome.

DETAILED DESCRIPTION:
Red blood cell transfusions are extremely common medical interventions, yet, it remains unclear when patients should be transfused. This pilot study will evaluate the feasibility of conducting a research protocol that will lead to a large scale clinical trial designed to evaluate the treatment effectiveness of two transfusion threshold strategies in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older;
* STEMI (ST segment elevated myocardial infarction)
* NSTEMI (Non ST segment elevation myocardial infarction)
* unstable angina
* stable coronary artery disease (undergoing cardiac catheterization during the index hospitalization);
* written informed consent has been obtained
* hemoglobin concentration less than 10 g/dL at the time of random allocation.

Exclusion Criteria:

* bleeding cannot be controlled at the cardiac catheterization puncture site and/or require surgery to repair vessel
* retroperitoneal bleeding requiring surgery
* clinically important hemodynamic instability based on the judgment of the treating physician
* terminal malignancy or life expectancy less than 6 months
* scheduled for cardiac surgery within the next 30 days
* symptomatic at the time of randomization
* declines blood transfusion
* history of a clinically significant transfusion reaction
* inability to provide informed consent;
* enrolled in a competing study
* previous participation in the MINT trial
* any patient who in the judgment of the research team should not be enrolled in the trial. This would include, but not be limited to, factors such alcohol or drug dependence, or psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Carson, MD, Study Chair — Rutgers, The State University of New Jersey; Sheryl F Kelsey, PhD, Principal Investigator — University of Pittsburgh Data Coordinating Center
Locations (7):
- United States (7):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Jack D. Weiler Hospital of Montefiore Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh Data Coordinating Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Result] Carson JL, Brooks MM, Abbott JD, Chaitman B, Kelsey SF, Triulzi DJ, Srinivas V, Menegus MA, Marroquin OC, Rao SV, Noveck H, Passano E, Hardison RM, Smitherman T, Vagaonescu T, Wimmer NJ, Williams DO. Liberal versus restrictive transfusion thresholds for patients with symptomatic coronary artery disease. Am Heart J. 2013 Jun;165(6):964-971.e1. doi: 10.1016/j.ahj.2013.03.001. Epub 2013 Apr 8. PMID 23708168
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Started | 55 | 55
Completed | 55 | 54
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (13.6) | 74.3 (11.1) | 70.8 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Concentration
Description: Differences in the mean hemoglobin concentrations between the two study arms.
Time Frame: In-hospital up to 30 days post randomization
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 55
g/dL
  Hemoglobin Day 1 Post Randomization | 10.30 (1.00) | 9.03 (0.82)
  Hemoglobin Day 2 Post Randomization | 10.78 (0.78) | 8.98 (0.80)
  Hemoglobin Day 3 Post Randomization | 10.64 (0.71) | 9.12 (0.75)
Statistical Analysis 1: Comparison: Liberal Transfusion Strategy vs Restrictive Transfusion Strategy; Day 1 Post Randomization; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Liberal Transfusion Strategy vs Restrictive Transfusion Strategy; Day 2 Post Randomization; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Liberal Transfusion Strategy vs Restrictive Transfusion Strategy; Day 3 Post Randomization; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Primary Outcome: Red Blood Cell Transfusion
Description: Differences in mean number of units of red blood cell transfusions between the two study arms.
Time Frame: In-hospital up to 30 days post randomization
Measure: Mean (Standard Deviation); unit: blood units
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 55
blood units | 1.58 (1.13) | 0.49 (1.03)
Statistical Analysis 1: Comparison: Liberal Transfusion Strategy vs Restrictive Transfusion Strategy; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Mortality or Myocardial Ischemia
Description: Composite 30 day rates of all cause 30 day mortality, or myocardial infarction (recurrent if had ST segment or Non ST segment MI or new myocardial infarction) up to 30 days after randomization, or unscheduled coronary revascularization within 30 days.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants | 6 | 14
Statistical Analysis 1: Comparison: Liberal Transfusion Strategy vs Restrictive Transfusion Strategy; Test type: Superiority or Other; Risk Ratio (RR) = 2.38, 95% CI 2-sided [0.99 to 5.73] — Restrictive Arm (numerator) compared to Liberal Arm (denominator)

4. Secondary Outcome: Mortality or Myocardial Ischemia
Description: Composite 6 month rates of all cause 6 month mortality, recurrent myocardial infarction up to 6 months after randomization, unscheduled coronary revascularization within 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants | 15 | 20
Statistical Analysis 1: Comparison: Liberal Transfusion Strategy vs Restrictive Transfusion Strategy; Test type: Superiority or Other; Risk Difference (RD) = 9.7, 95% CI [-5.3 to 24.7] — Restrictive Arm (numerator) compared to Liberal Arm (denominator)

5. Secondary Outcome: Individual Components of Composite Outcome
Description: All cause mortality Myocardial infarction (recurrent if had ST segment or Non ST segment MI or new myocardial infarction) Unscheduled coronary revascularization.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants
  Mortality | 1 | 7
  Myocardial Infarction | 5 | 7
  Unscheduled Coronary Revascularization | 0 | 2
Statistical Analysis 1: Comparison: Liberal Transfusion Strategy vs Restrictive Transfusion Strategy; Mortality; Test type: Superiority or Other; Risk Ratio (RR) = 7.13, 95% CI 2-sided [0.91 to 56.02] — Restrictive Arm (numerator) compared to Liberal Arm (denominator)
Statistical Analysis 2: Comparison: Liberal Transfusion Strategy; Myocardial Infarction; Test type: Superiority or Other; Risk Ratio (RR) = 1.43, 95% CI 2-sided [0.48 to 4.22] — Restrictive Arm (numerator) compared to Liberal Arm (denominator)

6. Secondary Outcome: Mortality From Cardiac Causes
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants | 1 | 7

7. Secondary Outcome: Unscheduled Hospital Admission
Description: Unscheduled hospital admission at 30 days for any reason, for cardiac reason (e.g., acute coronary syndrome, MI, congestive heart failure, or arrhythmia), or infection.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants
  Any Readmission | 9 | 17
  Cardiac Readmission | 3 | 8
  Infection Readmission | 0 | 2

8. Secondary Outcome: Stroke
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants | 1 | 0

9. Secondary Outcome: Congestive Heart Failure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants | 2 | 7

10. Secondary Outcome: Stent Thrombosis
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants | 0 | 0

11. Secondary Outcome: Deep Vein Thrombosis or Pulmonary Embolism
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants | 1 | 0

12. Secondary Outcome: Pneumonia or Blood Stream Infection and Each Separately
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants
  Pneumonia or Blood Stream Infection | 0 | 2
  Pneumonia | 0 | 2
  Blood Stream Infection | 0 | 0

13. Secondary Outcome: Composite Mortality and Morbidity
Description: Composite rates of all cause mortality, or myocardial infarction (recurrent if had ST segment or Non ST segment MI or new myocardial infarction), or unscheduled coronary revascularization or pneumonia.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 55 | 54
Participants | 6 | 16

ADVERSE EVENTS:
Time Frame: Up to 6 months following randomization
Description: Obtained via telephone follow-up and, if relevant, medical record review
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Serious Adverse Events (participants affected / at risk) | 7/55 | 10/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liberal Transfusion Strategy (N=55) | Restrictive Transfusion Strategy (N=54)
Death at 6 months (Cardiac disorders) | 7 (7) | 10 (10)
Myocardial Infarction at 30 days (Cardiac disorders) | 5 (5) | 7 (7)
Congestive Heart Failure at 30 Days (Cardiac disorders) | 2 (2) | 7 (7)

LIMITATIONS AND CAVEATS:
This pilot trial was not designed to enroll enough patients to answer the transfusion dilemma currently facing clinicians in practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes